CLINICAL TRIAL: NCT01154725
Title: Effect of Patient Education and Rehabilitational Interventions on Health Related Quality of Life of Patients With Permanent Stomas Regardless of Cause
Brief Title: The Effect of Patient Education and Rehabilitation on Quality of Life in Patients With Permanent Stomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Anne Kjærgaard Danielsen, Ph.d.student, RN, Herlev Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AKD01
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Colostomy
Keywords: Patient education; Health-Related Quality of Life; patients with stomas; stomatherapy; health economics
MeSH Terms: interventions — Patient Education as Topic; Rehabilitation; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Habitual stoma care (Other): habitual patient education
  Interventions: Behavioral: habitual patient education
- Patient education and rehabilitation (Experimental): patient education and rehabilitation
  Interventions: Behavioral: Patient education and rehabilitation

INTERVENTIONS:
Behavioral: Patient education and rehabilitation — Patients in the experimental group will receive specialized and optimized care by stoma care nurses. This includes one-on-one guiding during the hospitalization, guidance by telephone after discharge and participation in patient education 3 times after discharge.
  Other Names: health related quality of life; patient education; stoma care; stomatherapy; telephone guidance; group based learning
  Arms: Patient education and rehabilitation
Behavioral: habitual patient education — habitual patient education
  Arms: Habitual stoma care

SUMMARY:
The purpose of the experiment is to study the effect it has on patients' quality of life if they go through a structured process marked by intensified and specialized effort by ostomy nurse. This includes close monitoring during hospitalization, telephone contact and guidance following discharge and participation in a group based patient school up to 4 months after discharge .

At the same time the study also examines what the economic effect of following the intervention will have.

DETAILED DESCRIPTION:
Construction of an ostomy is a radical treatment with permanent physical signs of body alteration. It leads to loss of a central and very personal bodily function (excretion of faeces through the rectum) and there is a significant change in personal hygiene.

Having a colostomy is not a uniform state but is characterized by many different factors: Several types of ostomy, several underlying causes that lead to stoma creation such as cancer, several individual psychosocial profile, which naturally affect individuals differently. Patients are forced to living with a changed body image, a change in daily routines, and for some there will also be changes in lifestyle, social standing and their sexuality will be affected. At the same time patients experience a break when they are discharged from the hospital, and they may lack the practical and emotional support.

The training and education of patients is increasingly being carried out by stoma nurses both in Denmark and internationally. The primary role is to inform and prepare patients before surgery and to keep the contact with patients after surgery to ensure the fulfillment of the patient´s independent and meaningful life after ostomy construction. It is assumed that ostomy nurse's intervention and involvement are important for the patient's quality of life, but there are no studies that uniquely identifies the type of education that has the greatest effect, which applies both to content and methods.

Quality of life measurement in health care is a merging method to ensure the patient´s perspective on health treatments.It is greatly needed to test the efficacy of nursing interventions on patients' quality of life. Pressure on health services increase which makes it imperative also to include analysis and calculation of economic effect of the intervention.

ELIGIBILITY:
Inclusion criteria:

* All patients with permanent or temporary stomas regardless of cause that are expected to be able to cooperate in filling out questionnaires and who will participate in the planned interventions.

Exclusion criteria:

* Patients that post-operatively are not able to cooperate and participate in the planned interventions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-08; Primary Completion 2011-11 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Ostomy Adjustment Scale measurement of quality of life | 6 months (+/- 2 weeks) postoperatively
  the study measures quality of life both with the disease specific questionnaire Ostomy Adjustment Scale and also with a generic questionnaire Sf-36.

SECONDARY OUTCOMES:
Economic effect | 6 months after discharge
  The investigators will monitor readmittance and contacts and diagnostic procedures and therapeutic interventions related to stoma creation during the period from admittance to hospital until 6 months after discharge.
Ostomy Adjustment Scale and SF-36 measurement of quality of life | 3 months (+/-2 weeks) postoperatively
  the study measures quality of life both with the disease specific questionnaire Ostomy Adjustment Scale and also with a generic questionnaire Sf-36.
Ostomy Adjustment Scale and SF-36 measurement of quality of life | 3-7 days postoperatively before discharge
  the study measures quality of life both with the disease specific questionnaire Ostomy Adjustment Scale and also with a generic questionnaire Sf-36.
SF-36 measurement of quality of life | 6 months (+/- 2 weeks) postoperatively
  the study measures quality of life both with the disease specific questionnaire Ostomy Adjustment Scale and also with a generic questionnaire Sf-36.

CONTACTS AND LOCATIONS:
Overall Officials: Anne K Danielsen, Nurse, MaClN, Principal Investigator — Herlev University Hospital, Department of Gastroenterology
Locations (2):
- Denmark (2):
  - Department of Surgery, Herlev University Hospital, Herlev
  - Herlev University Hospital, Herlev

REFERENCES:
- [Derived] Danielsen AK, Rosenberg J. Patient education after stoma creation may reduce health-care costs. Dan Med J. 2014 Apr;61(4):A4659. PMID 24814582
- [Derived] Danielsen AK, Rosenberg J. Health related quality of life may increase when patients with a stoma attend patient education--a case-control study. PLoS One. 2014 Mar 7;9(3):e90354. doi: 10.1371/journal.pone.0090354. eCollection 2014. PMID 24609004